CLINICAL TRIAL: NCT00089583
Title: A 48 Week, Phase II, Non-Comparative, Open-label, Multi-Cohort, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of GW433908/Ritonavir BID When Administered to HIV-1 Infected, PI-Naïve and Experienced, Pediatric Subjects, 2 to 18 Years Old and of GW433908 BID Administered to PI-Naïve, Pediatric Subjects 2 to < 6 Years Old
Brief Title: 48-Week Study Of GW433908 And Ritonavir Or GW433908 Alone, Twice Daily In Pediatric Patients With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APV29005
Record Dates: First submitted 2004-08-06; First posted 2004-08-10 (Estimated); Results first posted 2012-06-21 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Infection, Human Immunodeficiency Virus I
Keywords: antiretroviral therapy; pediatrics; AGENERASE; amprenavir; fosamprenavir; HIV Infection; ritonavir; protease inhibitor; LEXIVA
MeSH Terms: conditions — Infections; HIV Infections | interventions — fosamprenavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 - 18 yrs old (FPV/RTV BID) (Experimental): Cohort 1B - 2 - less than 6yrs old (FPV/RTV BID) Cohort 2 - 6 to less than 12 yrs old (FPV/RTV BID) Cohort 3 - 12 - 18 yrs old (FPV/RTV BID) Cohort 4 - 2 - 18 yrs (FPV/RTV BID)
  Interventions: Drug: LEXIVA (GW433908); Drug: Ritonavir
- 2 - less than 6yrs old (FPV BID) (Experimental): Cohort 1A - 2 - less than 6yrs old (FPV BID)
  Interventions: Drug: LEXIVA (GW433908)

INTERVENTIONS:
Drug: LEXIVA (GW433908) — Fosamprenavir suspension or tablet bid
Drug: Ritonavir — Ritonavir solution bid
  Other Names: LEXIVA (GW433908)
  Arms: 2 - 18 yrs old (FPV/RTV BID)

SUMMARY:
This is a 48-week study to collect information on the safety and activity of an investigational medicine in patients, ages 2 to 18 years old, with HIV infection .

DETAILED DESCRIPTION:
A 48 Week, Phase II, non-comparative, open-label, multi-cohort, multicenter study to evaluate the safety, tolerability, pharmacokinetics and antiviral activity of GW433908/Ritonavir BID when administered to HIV-1 infected PI-Naive and experienced, Pediatric Subjects 2 to 18 years old and of GW433908 BID Administered to PI-Naive Pediatric subjects 2 to <6 years old

ELIGIBILITY:
Inclusion criteria:

* Males or females 2 to 18 years of age Cohorts 1A and 1B, up to one month before 6th birthday at Baseline/Day 1 Cohort 2, up to one month before 12th birthday at Baseline/Day 1 Cohort 3, up to one month before 19th birthday at Baseline/Day 1
* A female is eligible to enter and participate in this study if she is of:

  1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is pre-menarchial); or,
  2. child-bearing potential with a negative serum pregnancy test at screen, a negative urine pregnancy test on Day 1 and who agrees to use one of the following methods of contraception (any contraception method must be used consistently and correctly, i.e., in accordance with both the product label and the instructions of a physician). Premenarchial females who develop child-bearing potential while on the study will be expected to follow one of the methods of contraception listed below.

Agreement for complete abstinence from intercourse from 2 weeks prior to administration of study drugs, throughout the study and for 2 weeks after discontinuation of all study medications. Should a female subject of childbearing potential decide to become sexually active during the course of the study, she must be counseled and be willing to use one of the contraception methods listed below:

Double barrier contraception (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide) Any intrauterine device (IUD) with published data showing that the expected failure rate is less than 1% per year (not all IUDs meet this criterion) Any other method with published data showing that the lowest expected failure rate for that method is less than 1% per year.

Hormonal contraception is not recommended, due to decreased efficacy of contraception as well as increased risk of hepatic transaminase elevation (see Section 8.2).

All subjects of childbearing potential or developing child-bearing potential while participating in this study should be counseled on the practice of safe/safer sex.

* Parent or legal guardian (and subject whenever possible) has the ability to understand and provide written informed consent for the subject to participate in the trial. Verbal witnessed assent must be obtained from the subject whenever possible.
* Screening plasma HIV-1 RNA >=400copies/mL.
* Subjects must meet one of the following criterion:

Antiretroviral therapy (ART)-naïve or PI-naïve subjects (defined as having received less than one week of any PI and any length of therapy with Nucleoside Reverse Transcriptase Inhibitors (NRTIs) and/or Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs)).

PI-experienced subjects (defined as having received greater than one week prior PI therapy with no more than three PIs). Prior RTV boosted PI therapy will be considered as only one PI as long as the RTV dose was lower than that recommended for use of RTV as an antiretroviral age

Exclusion criteria:

* Prior history of having received APV or FPV for >7 days.
* NNRTI use within 14 days prior to study drug administration or anticipated need for concurrent NNRTI therapy during the treatment period of the study.
* Subjects who, in the investigator's opinion, are not able to comply with the requirements of the study.
* Subject is in the initial acute phase of a Centers for Disease Control and Prevention (CDC) Clinical Category C event or infection (per 1994 classification) at Baseline. Subject may be enrolled provided they are receiving treatment for the infection, such treatment not being contraindicated with FPV, and the subjects are clinically improving at the Baseline visit.
* Presence of a malabsorption syndrome or other gastrointestinal dysfunction which might interfere with drug absorption or render the subject unable to take oral medication.
* Pregnant or lactating females.
* Presence of any serious medical condition (e.g., hemoglobinopathy, chronic anemia, a history of insulin resistance, diabetes, cardiac dysfunction, hepatitis or clinically relevant pancreatitis) which, in the opinion of the investigator, might compromise the safety of the subject.
* Grade 3 or 4 transaminase levels (ALT and/or AST) within 28 days prior to study drug administration and/or clinically relevant episodes of hepatitis within the previous 6 months.
* Any acute laboratory abnormality at screen which, in the opinion of the investigator, should preclude the subject's participation in the study of an investigational compound. If subjects are found to have an acute Grade 4 laboratory abnormality at screening, this test may be repeated once within the screening window. Any verified Grade 4 laboratory abnormality at screen would exclude a subject from study participation.
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days of study drug administration or an anticipated need for such treatment within the study period.
* Treatment with immunomodulating agents (e.g., systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (e.g., hydroxyurea or foscarnet) within 28 days of study drug administration.
* Treatment with any of the following medications within 28 days prior to receiving study medication or the anticipated need during the study:

Drugs whose plasma concentration may be increased to unsafe levels when co-administered with FPV including:

Amiodarone, astemizole, bepridil, cisapride, dihydroergotamine, ergonovine, ergotamine, flecainide, halofantrine, lidocaine, lovastatin, methylergonovine, midazolam, pimozide, propafenone, quinidine, simvastatin, terfenadine, and triazolam

Drugs with the potential to significantly decrease plasma APV concentrations including:

Carbamazepine, dexamethasone, phenobarbital, primidone, rifampin, St Johns Wort.

* Treatment with other investigational drugs/therapies (note: treatments available through a Treatment Investigational New Drug [IND] or other expanded-access mechanism will be evaluated on a case-by-case basis in consultation with the sponsor) within 28 days prior to study drug administration or during the treatment period of the study.
* History of drug or other allergy which, in the opinion of the investigator, contraindicates participation in the trial or known hypersensitivity to any study medications (e.g., documented hypersensitivity to a nucleoside analogue).
* Substantial non-adherence based on history

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2004-07; Primary Completion 2011-03 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (32):
- United States (13):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
- GSK Investigational Site, Antwerp, Belgium
- Canada (4):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Bucharest, Romania
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Africa (4):
  - GSK Investigational Site, Coronationville, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Parow Valley, Western Province
  - GSK Investigational Site, Soweto
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo ( Pontevedra)

REFERENCES:
- [Background] Voronin E, Fortuny C, Perez-Tamarit D, et al. Pharmacokinetics, safety and antiviral activity of fosamprenavir-containing regimens in HIV-infected 2 to 18 year-old children (48-week data, Study APV29005, a prospective, open-label, multi-centre, 48-week cohort study). Presented at: AIDS 2012 - 19th International AIDS Conference; July 22-27, 2012; Washington, DC.
- [Background] Ross L, Cotton M, Cassim H, et al. HIV-1 drug resistance and mutational profile in fosamprenavir-treated HIV-infected children aged 2 months to 18 years at start of therapy. Presented at: AIDS 2012 - 19th International AIDS Conference; July 22-27, 2012; Washington DC.
- [Result] Fortuny C, Duiculescu D, Cheng K, Garges HP, Cotton M, Tamarirt DP, Ford SL, Wire MB, Givens N, Ross LL, Lou Y, Perger T, Sievers J. Pharmacokinetics and 48-week safety and antiviral activity of fosamprenavir-containing regimens in HIV-infected 2- to 18-year-old children. Pediatr Infect Dis J. 2014 Jan;33(1):50-6. doi: 10.1097/INF.0b013e3182a1126a. PMID 23811744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 110 participants (par.) were enrolled in the study; however, 1 par. withdrew from the study prior to the first dose of study drug and was not included in the Intent-to-Treat Exposed or Safety Populations. Therefore, 109 par. received >=1 dose of study drug and are thus categorized as starting the study in the Participant Flow module.
Groups:
- FPV Treatment Group: Human immunodeficiency virus type 1 (HIV-1)-infected, protease inhibitor (PI)-naïve pediatric participants, 2 to <6 years old, receiving fosamprenavir (FPV) oral suspension 30-40 milligrams per kilogram (mg/kg) twice a day (BID). PI-naïve participants are defined as those participants who received less than one week of any PI and any length of therapy with nucleoside reverse transcriptase inhibitors (NRTIs) and/or non-NRTIs (NNRTIs).
- FPV/RTV Treatment Group: HIV-1-infected, PI-naïve and -experienced pediatric participants, 2 to 18 years old, receiving FPV boosted with ritonavir (FPV/RTV) BID. Participants who were 2-<6 years old received FPV oral suspension/ritonavir oral solution 20/4 or 23/3 mg/kg BID; participants who were 6 years old or older received FPV oral suspension/RTV oral solution 15/3 or 18/3 mg/kg BID. A 700/100 mg BID tablet regimen was administered to participants able to take tablets/capsules. PI-experienced participants are defined as those participants who received more than one week of prior PI therapy with no more than three PIs. Prior RTV-boosted therapy was considered as only one PI as long as the RTV dose was lower than that recommended for use of RTV as an antiretroviral agent.
Period: Overall Study
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Started | 20 | 89
Completed | 13 | 51
Not Completed | 7 | 38
Not completed — Adverse Event | 0 | 3
Not completed — Insufficient Viral Load Response | 5 | 5
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Participant (Par) Didn't Take Medication | 1 | 0
Not completed — Participant Refused Study Medication | 0 | 2
Not completed — Non-Compliance | 0 | 4
Not completed — Poor Medical Compliance/Adherence Issues | 0 | 3
Not completed — Participant Management Criteria Met | 0 | 1
Not completed — Reason Not Provided | 0 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Principal Investigator Decision | 0 | 10
Not completed — Start of Disallowed Medication | 0 | 1
Not completed — Necessity to Use Prohibited Drug | 1 | 0
Not completed — Participant Incarcerated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group | Total
Number analyzed (Participants) | 20 | 89 | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 2.9 (1.07) | 10.0 (4.49) | 8.7 (4.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 43 | 58
  Male | 5 | 46 | 51
Race/Ethnicity, Customized [Number; unit: participants]
  Arabic/North African | 0 | 1 | 1
  Black | 0 | 43 | 43
  South Asian | 0 | 1 | 1
  White/Caucasian | 19 | 41 | 60
  Race Not Specified | 1 | 3 | 4
Par with the Indicated 1993 Center for Disease Control and Prevention (CDC) Baseline Classification [Number; unit: participants] — The adult/adolescent (>=13 years) HIV infection CDC classification system was based on 3 categories (Cat). Cat A, asymptomatic acute/primary HIV infection or persistent generalized lymphadenopathy. Cat B, symptomatic conditions not included in Cat A or C but attributed to a cell-mediated immunity defect or for which the clinical course or management was complicated by HIV infection. Cat C, acquired immune deficiency syndrome (AIDS)-defining conditions. Infected children (<13 years) are classified into mutually exclusive categories per 3 parameters: infection, clinical, and immunologic status.
  participants
    <13 years (yrs); mildly symptomatic (S) | 18 | 26 | 44
    <13 yrs; moderately S | 1 | 15 | 16
    <13 yrs; severely S | 0 | 10 | 10
    <13 yrs; non-S | 1 | 5 | 6
    >=13 yrs; asymptomatic/lymphadenopathy/acute HIV | 0 | 12 | 12
    >=13 yrs; asymptomatic, not AIDS | 0 | 14 | 14
    >=13 yrs; AIDS | 0 | 5 | 5
    >=13 yrs; not reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Plasma Amprenavir (APV) AUC (0-tau[τ])
Description: Plasma samples were assayed for APV concentrations using a validated assay. The GlaxoSmithKline (GSK) Department of Clinical Pharmacology Modeling and Simulation conducted pharmacokinetic (PK) analysis of the plasma APV concentration-time data using a model-independent approach. As a measure of total drug exposure, the area under the plasma-concentration-versus-time curve over the dosing interval at steady-state (AUC[0-τ]), where τ is the length of the dosing interval, was calculated by the linear up/log down trapezoidal method. hr, hour; µg, micrograms; mL, milliliter.
Time Frame: Week 48
Population: Pharmacokinetic (PK) Population: all participants for whom serial plasma PK samples were analyzed. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*µg/mL
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 9 | 14
hr*µg/mL
  2 to <6 yrs, 30 mg/kg BID; n=9, 0 | 22.3 [15.3 to 32.6] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6 yrs, 40 mg/kg BID; n=7, 0 | 24.1 [15.2 to 38.0] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6 yrs, 23/3 mg/kg BID; n=0, 14 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 55.3 [37.9 to 80.7]
  6 to <12 yrs, 15/3 mg/kg BID; n=0, 9 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 32.3 [23.0 to 45.3]
  6 to <12 yrs, 18/3 mg/kg BID; n=0, 12 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 48.4 [38.1 to 61.4]
  6 to <12 yrs, 700/100 mg BID; n=0, 3 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 37.6 [22.2 to 63.8]
  12 to 18 yrs, 15/3 mg/kg BID; n=0, 4 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 21.8 [18.0 to 26.3]
  12 to 18 yrs, 18/3 mg BID; n=0, 3 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 41.7 [16.2 to 108]
  12 to 18 yrs, 700/100 mg BID; n=0, 13 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 35.3 [28.2 to 44.1]

2. Primary Outcome: Plasma APV Cmax
Description: The maximum concentration at steady state (Cmax) was measured.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter (µg/mL)
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 9 | 14
Micrograms per milliliter (µg/mL)
  2 to <6 yrs, 30 mg/kg BID; n=9, 0 | 7.15 [5.05 to 10.10] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6 yrs, 40 mg/kg BID; n=7, 0 | 6.52 [4.47 to 9.51] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6 yrs, 23/3 mg/kg BID; n=0, 14 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 8.66 [6.08 to 12.30]
  6 to <12 yrs, 15/3 mg/kg BID; n=0, 10 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 4.34 [3.16 to 5.96]
  6 to <12.yrs, 18/3 mg/kg BID; n=0, 12 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 6.40 [5.02 to 8.15]
  6 to <12 yrs, 700/100 mg BID; n=0, 3 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 5.85 [3.94 to 8.70]
  12 to 18 yrs, 15/3 mg/kg BID; n=0, 4 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 3.92 [2.44 to 6.29]
  12 to 18 yrs, 18/3 mg/kg BID; n=0, 4 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 4.91 [2.69 to 8.97]
  12 to 18 yrs, 700/100 mg BID; n=0, 13 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 4.93 [3.83 to 6.34]

3. Primary Outcome: Plasma APV Cτ
Description: The plasma concentration at the end of the dosing interval at steady-state (Cτ) was measured.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter (µg/mL)
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 19 | 40
Micrograms per milliliter (µg/mL)
  2 to <6 yrs, 30 mg/kg BID; n=19, 0 | 0.55 [0.41 to 0.75] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6 yrs, 40 mg/kg BID; n=10, 0 | 0.70 [0.41 to 1.19] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6 yrs, 23/3 mg/kg BID; n=0, 16 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 3.39 [2.51 to 4.57]
  6 to <12 yrs, 15/3 mg/kg BID; n=0, 13 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 2.24 [1.70 to 2.93]
  6 to <12 yrs, 18/3 mg/kg BID; n=0, 23 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 2.42 [1.90 to 3.07]
  6 to <12 yrs, 700/100 mg BID; n=0, 7 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 1.81 [0.80 to 4.08]
  12 to 18 yrs, 15/3 mg/kg BID; n=0, 6 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 1.45 [0.56 to 3.74]
  12 to 18 yrs, 18/3 mg/kg BID; n=0, 10 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 1.80 [1.22 to 2.67]
  12 to 18 yrs, 700/100 mg BID; n=0, 40 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 2.01 [1.74 to 2.32]

4. Primary Outcome: Plasma APV CL/F Following Dosing Expressed in mg/kg
Description: Apparent clearance of drug from plasma following extravascular administration (CL/F) was calculated using the formulation: APV Dose in mg/kg units divided by AUC(0-τ). For FPV, doses were expressed in APV molar equivalents (50 mg of FPV = 43.2 mg of APV). Normalizing CL/F for bodyweight allows for comparison of CL/F across populations.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters/minute/kilogram (mL/min/kg)
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 9 | 14
Milliliters/minute/kilogram (mL/min/kg)
  2 to <6yrs, 30 mg/kg BID; n=9, 0 | 19.3 [13.2 to 28.2] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6yrs, 40 mg/kg BID; n=7, 0 | 23.4 [14.9 to 36.8] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6yrs, 23/3 mg/kg BID; n=0, 14 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 6.06 [4.12 to 8.91]
  6 to <12 yrs, 15/3 mg/kg BID; n=0, 9 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 6.48 [4.68 to 8.98]
  6 to <12 yrs, 18/3 mg/kg BID; n=0, 12 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 5.27 [4.16 to 6.68]
  6 to <12 yrs, 700/100 mg BID; n=0, 3 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 5.94 [2.59 to 13.9]
  12 to 18 yrs, 15/3 mg/kg BID; n=0, 4 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 10.1 [8.35 to 12.3]
  12 to 18 yrs, 18/3 mg BID; n=0, 3 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 6.00 [2.37 to 15.2]
  12 to 18 yrs, 700/100 mg BID; n=0, 13 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 5.33 [4.26 to 6.68]

5. Primary Outcome: Plasma APV CL/F Following Dosing Expressed in mg
Description: Apparent clearance of drug from plasma following extravascular administration (CL/F) was calculated as dose/AUC(0-τ). For FPV, doses were expressed in APV molar equivalents (50 mg of FPV = 43.2 mg of APV).
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters per minute (mL/min)
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 9 | 14
Milliliters per minute (mL/min)
  2 to <6yrs, 30 mg/kg BID; n=9, 0 | 269 [193 to 376] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6yrs, 40 mg/kg BID; n=7, 0 | 330 [203 to 538] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6yrs, 23/3 mg/kg BID; n=0, 14 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 91 [60 to 139]
  6 to <12 yrs, 15/3 mg/kg BID; n=0, 9 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 195 [136 to 279]
  6 to <12 yrs, 18/3 mg/kg BID; n=0, 12 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 149 [104 to 214]
  6 to <12 yrs, 700/100 mg BID; n=0, 3 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 266 [157 to 452]
  12 to 18 yrs, 15/3 mg/kg BID; n=0, 4 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 392 [355 to 432]
  12 to 18 yrs, 18/3 mg BID; n=0, 3 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 198 [47 to 838]
  12 to 18 yrs, 700/100 mg BID; n=0, 13 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 284 [227 to 354]

6. Primary Outcome: Plasma APV Tmax
Description: The time to reach the maximum concentration (Cmax) at steady state is defined as tmax.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 9 | 14
hours
  2 to <6yrs, 30 mg/kg BID; n=9, 0 | 1.17 [1.00 to 3.75] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6yrs, 40 mg/kg BID; n=7, 0 | 1.00 [0.75 to 2.00] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6yrs, 23/3 mg/kg BID; n=0, 14 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 1.25 [1.00 to 4.00]
  6 to <12 yrs, 15/3 mg/kg BID; n=0, 10 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 2.00 [1.00 to 6.00]
  6 to <12 yrs, 18/3 mg/kg BID; n=0, 12 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 1.96 [0.50 to 4.00]
  6 to <12 yrs, 700/100 mg BID; n=0, 3 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 3.92 [1.00 to 4.02]
  12 to 18 yrs, 15/3 mg/kg BID; n=0, 4 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 1.00 [1.00 to 2.00]
  12 to 18 yrs, 18/3 mg BID; n=0, 3 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 1.50 [0.00 to 2.00]
  12 to 18 yrs, 700/100 mg BID; n=0, 13 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 2.00 [0.92 to 7.97]

7. Primary Outcome: Plasma APV t1/2
Description: The apparent terminal phase half-life (t1/2) is calculated as loge2/λz. The apparent terminal phase rate constant (λz) is the slope of the terminal portion of the logarithmically transformed concentration-time data as estimated by linear regression.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 9 | 14
hours
  2 to <6yrs, 30 mg/kg BID; n=9, 0 | 3.03 [2.09 to 4.41] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6yrs, 40 mg/kg BID; n=5, 0 | 3.18 [2.14 to 4.73] | NA [NA to NA] — No participants were analyzed at this dose in this age group.
  2 to <6yrs, 23/3 mg/kg BID; n=0, 14 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 5.21 [4.47 to 6.08]
  6 to <12 yrs, 15/3 mg/kg BID; n=0, 7 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 10.5 [8.36 to 13.1]
  6 to <12 yrs, 18/3 mg/kg BID; n=0, 10 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 8.41 [5.90 to 12.0]
  6 to <12 yrs, 700/100 mg BID; n=0, 2 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 7.43 [NA to NA] — When n<=2, 95% CI data will not be provided.
  12 to 18 yrs, 15/3 mg/kg BID; n=0, 4 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 6.12 [3.67 to 10.2]
  12 to 18 yrs, 18/3 mg BID; n=0, 4 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 8.76 [2.79 to 27.5]
  12 to 18 yrs, 700/100 mg BID; n=0, 11 | NA [NA to NA] — No participants were analyzed at this dose in this age group. | 7.64 [4.84 to 12.0]

8. Primary Outcome: Number of Participants Who Permanently Discontinued the Treatment Due to Any Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Week 48
Population: Safety Population: all participants with documented evidence of having received at least one dose of investigational treatment.
Measure: Number; unit: participants
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 20 | 89
participants | 0 | 4

9. Primary Outcome: Change From Baseline in Triglycerides, Total Cholesterol, Low-density Lipoprotein (LDL) Cholesterol, High-density Lipoprotein (HDL) Cholesterol, and Serum Glucose at Week 48
Description: Blood samples of all participants were collected under fasting conditions for the evaluation of triglycerides, total cholesterol, HDL cholesterol, LDL cholesterol, and serum glucose. Clinical chemistry analyses were carried out using the observed analysis strategy. Change from Baseline in triglycerides, total cholesterol, HDL cholesterol, LDL cholesterol, and serum glucose was calculated as the value at Week 48 minus the value at Baseline.
Time Frame: Baseline (Day 1) and Week 48
Population: Safety Population. Only those participants contributing data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Millimoles per liter (mmol/L)
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 18 | 69
Millimoles per liter (mmol/L)
  Triglycerides; n=17, 65 | 0.1 [-0.2 to 0.3] | 0.2 [0.0 to 0.8]
  Total cholesterol; n=17, 65 | 1.1 [0.8 to 1.5] | 0.9 [0.2 to 1.6]
  HDL cholesterol; n=17, 65 | 0.4 [0.3 to 0.7] | 0.3 [0.1 to 0.4]
  LDL cholesterol; n=17, 64 | 0.6 [0.3 to 1.0] | 0.5 [-0.1 to 1.1]
  Glucose; n=18, 69 | 0.0 [-0.3 to 0.6] | 0.1 [-0.3 to 0.5]

10. Primary Outcome: Change From Baseline in Serum Lipase at Week 48
Description: Blood samples of all participants were collected for the evaluation of serum lipase. Clinical chemistry analyses were carried out using the observed analysis strategy. Change from Baseline in serum lipase was calculated as the value at Week 48 minus the value at Baseline.
Time Frame: Baseline (Day 1) and Week 48
Population: Safety Population. Only those participants contributing data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Units per liter (U/L)
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 18 | 69
Units per liter (U/L) | -2.0 [-5.0 to 0.0] | -1.0 [-7.0 to 4.0]

11. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) at Week 48
Description: Blood samples of the participants were collected for the evaluation of AST and ALT. Clinical chemistry analyses were carried out using the observed analysis strategy. Change from Baseline in AST and ALT was calculated as the value at Week 48 minus the value at Baseline.
Time Frame: Baseline (Day 1) and Week 48
Population: Safety Population. Only those participants contributing data were analyzed.
Measure: Median (Inter-Quartile Range); unit: International units per liter (IU/L)
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 18 | 70
International units per liter (IU/L)
  ALT | -3 [-14 to 19] | -7 [-16 to -1]
  AST | -6 [-19 to 10] | -9 [-17 to -4]

12. Primary Outcome: Number of Participants With Treatment-emergent (TE) Grade 3/4 Clinical Chemistry Laboratory Abnormalities
Description: A toxicity was considered TE if it was > than the Baseline grade, and if it was observed on/after the date of the first dose of study drug (SD), and on/before the date of the last dose of SD. Leucopenia is the decrease in the number of leucocytes (white blood cells [WBCs]); neutropenia is the decrease in the number of neutrophils (type of WBCs). Per the Division of AIDS Table for Grading the Severity of Adult and Pediatric AEs: Grade 3 is "severe"; Grade 4 is "potentially life-threatening." ULN, upper limit of normal; LDL, low-density lipoprotein; PC, platelet count.
Time Frame: Baseline (Day 1) until Week 48
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 20 | 87
participants
  ALT increased (inc.) (>5.0x ULN); n=20, 87 | 2 | 2
  AST inc. (>5.0x ULN); n=20, 87 | 2 | 2
  Cholesterol (Chol.) inc. (>7.77 mmol/L); n=16, 43 | 0 | 2
  Hyperglycemia (>13.88 mmol/L); n=16, 58 | 0 | 0
  Hypoglycemia (<2.22 mmol/L); n=16, 58 | 0 | 0
  LDL Chol. inc. (>=4.91 mmol/L); n=16, 43 | 0 | 4
  Triglycerides inc. (>8.48 mmol/L); n=16, 43 | 0 | 0
  Lipase inc. (>3.0x ULN); n=19, 85 | 0 | 0
  Leucopenia (<1.500 x 10^9/L); n=20, 84 | 0 | 0
  Neutropenia (<0.750 x 10^9/L); n=20, 84 | 8 | 7
  Hemoglobin > anemia (<1.16 mmol/L); n=20, 85 | 0 | 0
  PC > thrombocytopenia (<50.000 x 10^9/L); n=20, 85 | 0 | 1

13. Secondary Outcome: Plasma Ritonavir (RTV) AUC (0-τ)
Description: Plasma samples were assayed for RTV concentrations using a validated assay. The GlaxoSmithKline (GSK) Department of Clinical Pharmacology Modeling and Simulation conducted pharmacokinetic (PK) analysis of the plasma RTV concentration-time data using a model-independent approach. As a measure of total drug exposure, the area under the plasma-concentration-versus-time curve over the dosing interval at steady-state (AUC[0-τ]), where τ is the length of the dosing interval, was calculated by the linear up/log down trapezoidal method.
Time Frame: Week 48
Population: PK Population: all participants for whom a plasma PK sample was analyzed. Participants in the FPV arm did not take RTV; hence, they were not analyzed for this outcome measure. In the FPV/RTV arm, only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*µg/mL
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 15
hr*µg/mL
  2 to <6 yrs, 3 mg/kg BID; n=0, 10 |  | 3.98 [2.28 to 6.94]
  6 to <12 yrs, 3 mg/kg BID; n=0, 12 |  | 7.13 [5.37 to 9.46]
  6 to <12 yrs, 100 mg BID; n=0, 6 |  | 6.46 [3.60 to 11.6]
  12 to 18 yrs, 3 mg/kg BID; n=0, 1 |  | 5.74 [NA to NA] — Only one participant was analyzed at this dose in this age group.
  12 to 18 yrs, 100 mg BID; n=0, 15 |  | 6.13 [3.97 to 9.47]

14. Secondary Outcome: Plasma RTV Cmax
Description: The maximum concentration at steady state (Cmax) was measured.
Time Frame: Week 48
Population: PK Population. Participants in the FPV arm did not take RTV; hence, they were not analyzed for this outcome measure. In the FPV/RTV arm, only those participants contributing data at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 16
µg/mL
  2 to <6 yrs, 3 mg/kg BID; n=0, 10 |  | 0.633 [0.341 to 1.18]
  6 to <12 yrs, 3 mg/kg BID; n=0, 14 |  | 1.100 [0.779 to 1.54]
  6 to <12.yrs, 100 mg BID; n=0, 6 |  | 0.980 [0.572 to 1.68]
  12 to 18 yrs, 3 mg/kg BID; n=0, 3 |  | 0.750 [0.203 to 2.78]
  12 to 18 yrs, 100 mg BID; n=0, 16 |  | 1.06 [0.679 to 1.67]

15. Secondary Outcome: Plasma RTV Cτ
Description: The plasma concentration at the end of the dosing interval at steady-state (Cτ) was measured.
Time Frame: Week 48
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 41
µg/mL
  2 to <6 yrs, 3 mg/kg BID; n=0, 16 |  | 0.224 [0.179 to 0.279]
  6 to <12 yrs, 3 mg/kg BID; n=0, 24 |  | 0.297 [0.227 to 0.388]
  6 to <12 yrs, 100 mg BID; n=0, 10 |  | 0.228 [0.103 to 0.507]
  12 to 18 yrs, 3 mg/kg BID; n=0, 6 |  | 0.263 [0.135 to 0.510]
  12 to 18 yrs, 100 mg BID; n=0, 41 |  | 0.220 [0.177 to 0.273]

16. Secondary Outcome: Plasma RTV CL/F Following Dosing Expressed in mg/kg
Description: Apparent clearance of drug from plasma following extravascular administration (CL/F) was calculated using the formulation: RTV Dose in mg/kg units divided by AUC(0-τ). Normalizing CL/F for bodyweight allows for comparison of CL/F across populations.
Time Frame: Week 48
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min/kg
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 15
mL/min/kg
  2 to <6yrs, 3 mg/kg BID; n=0, 10 |  | 12.9 [7.33 to 22.7]
  6 to <12 yrs, 3 mg/kg BID; n=0, 12 |  | 6.81 [5.14 to 9.04]
  6 to <12 yrs, 100 mg/kg BID; n=0, 12 |  | 5.94 [3.56 to 9.94]
  12 to 18 yrs, 3 mg/kg BID; n=0, 1 |  | 8.61 [NA to NA] — Only one participant was analyzed at this dose in this age group.
  12 to 18 yrs, 100 mg BID; n=0, 15 |  | 5.59 [3.90 to 8.01]

17. Secondary Outcome: Plasma RTV CL/F Following Dosing Expressed in mg
Description: Apparent clearance of drug from plasma following extravascular administration (CL/F) was calculated as dose/AUC(0-τ).
Time Frame: Week 48
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 15
mL/min
  2 to <6yrs, 3 mg/kg BID; n=0, 10 |  | 195 [108 to 353]
  6 to <12 yrs, 3 mg/kg BID; n=0, 12 |  | 190 [142 to 253]
  6 to <12 yrs, 100 mg/kg BID; n=0, 6 |  | 258 [144 to 463]
  12 to 18 yrs, 3 mg/kg BID; n=0, 1 |  | 279 [NA to NA] — Only one participant was analyzed at this dose in this age group.
  12 to 18 yrs, 100 mg BID; n=0, 15 |  | 272 [176 to 420]

18. Secondary Outcome: Plasma RTV Tmax
Description: The time to reach the maximum concentration (Cmax) at steady state is defined as (tmax).
Time Frame: Week 48
Population: PK Population: all participants for whom a plasma PK sample was analyzed. Participants in the FPV arm did not take RTV; hence, they were not analyzed for this outcome measure. In the FPV/RTV arm, only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 15
hours
  2 to <6 yrs, 3 mg/kg BID; n=0, 10 |  | 3.92 [1.00 to 4.07]
  6 to <12 yrs, 3 mg/kg BID; n=0, 14 |  | 4.00 [0.50 to 11.92]
  6 to <12 yrs, 100 mg BID; n=0, 6 |  | 4.01 [1.00 to 11.92]
  12 to 18 yrs, 3 mg/kg BID; n=0, 3 |  | 5.92 [2.03 to 6.00]
  12 to 18 yrs, 100 mg BID; n=0, 16 |  | 3.96 [0.92 to 6.00]

19. Secondary Outcome: Plasma RTV t1/2
Description: alf-life (t1/2) is calculated as loge2/λz. The apparent terminal phase rate constant (λz) is the slope of the terminal portion of the logarithmically transformed concentration-time data as estimated by linear regression.
Time Frame: Week 48
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 14
hours
  2 to <6 yrs, 3 mg/kg BID; n=0, 10 |  | 3.43 [2.61 to 4.51]
  6 to <12 yrs, 3 mg/kg BID; n=0, 11 |  | 3.39 [2.88 to 4.00]
  6 to <12 yrs, 100 mg BID; n=0, 5 |  | 3.97 [3.17 to 4.97]
  12 to 18 yrs, 3 mg/kg BID; n=0, 1 |  | 2.84 [NA to NA] — Only one participant was analyzed at this dose in this age group.
  12 to 18 yrs, 100 mg BID; n=0, 14 |  | 3.64 [3.09 to 4.29]

20. Secondary Outcome: Plasma FPV AUC (0-τ)
Description: The majority of the FPV data were below the quantification limit. Therefore, plasma FPV PK parameters were not estimated.
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Plasma FPV Cmax and Cτ
Description: as for outcome 20
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Plasma FPV CL/F Following Dosing Expressed in mg/kg
Description: as for outcome 20
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Plasma FPV CL/F Following Dosing Expressed in mg
Description: as for outcome 20
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Plasma FPV Tmax
Description: as for outcome 20
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Plasma FPV t1/2
Description: as for outcome 20
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Number of Participants (Par.) With Virological Outcome (Plasma HIV-1 Ribonucleic Acid [RNA] <400 Copies/mL) at Week 48
Description: Blood samples of participants were collected to measure plasma HIV-1 RNA concentrations. PI-exp = PI-experienced.Virologic success was defined as plasma HIV-1 RNA <400 copies/mL. Virologic failure: (1) HIV-1 RNA >=400 copies/mL, (2) change of background antiretroviral treatment (ART), (3) discontinued study due to lack of efficacy, (4) discontinued study with last HIV-1 >=400 copies/mL. No virologic data at Week 48 window: (a) discontinued study due to an adverse event or death, (b) discontinued study due to other reasons, (c) missing data during window but still on study.
Time Frame: Week 48
Population: Intent-to-Treat Exposed (ITT-E) Population: par. with documented evidence of receiving >=1 treatment dose. Only par. contributing data were analyzed. The number of par. analyzed is the sum of the PI-naïve (received <1week's treatment with a PI) and -experienced (received >1week prior PI therapy with no more than 3 PIs before trial enrollment) par.
Measure: Number; unit: participants
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 20 | 89
participants
  PI-naïve, virological (V) success; n=20, 49 | 12 | 36
  PI-exp, V success; n=0, 40 | NA — No participants were analyzed for this population at this time point. | 19
  PI-naïve, V failure (1); n=20, 49 | 4 | 3
  PI-exp, V failure (1); n=0, 40 | NA — No participants were analyzed for this population at this time point. | 8
  PI-naïve, V failure (2); n=20, 49 | 2 | 4
  PI-exp, V failure (2); n=0, 40 | NA — No participants were analyzed for this population at this time point. | 7
  PI-naïve, V failure (3); n=20, 49 | 1 | 0
  PI-exp, V failure (3); n=0, 40 | NA — No participants were analyzed for this population at this time point. | 0
  PI-naïve;, V failure (4); n=20, 49 | 1 | 3
  PI-exp, V failure (4); n=0, 40 | NA — No participants were analyzed for this population at this time point. | 3
  PI-naïve, No V data at Week 48 (a); n=20, 49 | 0 | 1
  PI-exp, No V data at Week 48 (a); n=0, 40 | NA — No participants were analyzed for this population at this time point. | 1
  PI-naïve, No V data Week 48 (b); n=20, 49 | 0 | 1
  PI-exp, No V data at Week 48 (b); n=0, 40 | NA — No participants were analyzed for this population at this time point. | 0
  PI-naïve, No V data at Week 48 (c); n=20, 49 | 0 | 1
  PI-exp, No V data at Week 48 (c); n=0, 40 | NA — No participants were analyzed for this population at this time point. | 2

27. Secondary Outcome: Number of Participants (Par.) With Plasma HIV-1 Ribonucleic Acid (RNA) <400 Copies Per Milliliter at Baseline and Weeks 2,12, 24, and 48 (MSD=F)
Description: Blood samples of participants were collected to measure plasma HIV-1 RNA concentrations. PI-exp = PI-experienced. Viral load, measured in RNA copies per milliliter of plasma, is an efficacy measure for antiretroviral drugs. In the Missing, Switch, or Discontinuation = Failure (MSD=F) analysis, participants who had missing data at or had discontinued the study prior to a certain time point or had changed their background antiretroviral regimen are classified as non-responders.
Time Frame: Baseline and Weeks 2, 12, 24, and 48
Population: Intent-to-Treat Exposed (ITT-E) Population. Only those par. contributing data at the indicated time points were analyzed. The number of par. analyzed represents the sum of the PI-naïve (received <1 week's treatment with a PI) and -experienced (received >1week prior PI therapy with no more than 3 PIs before trial enrollment) par.
Measure: Number; unit: participants
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 20 | 89
participants
  PI-naïve, Baseline; n=20, 49 | 0 | 0
  PI-exp, Baseline; n=0, 40 | NA — No participants were analyzed for this population at this time point. | 0
  PI-naïve, Week 2; n=20, 49 | 3 | 9
  PI-exp, Week 2; n=0, 40 | NA — No participants were analyzed for this population at this time point. | 5
  PI-naïve, Week 12; n=20, 49 | 13 | 35
  PI-exp, Week 12; n=0, 40 | NA — No participants were analyzed for this population at this time point. | 19
  PI-naïve, Week 24; n=20, 49 | 13 | 35
  PI-exp, Week 24; n=0, 40 | NA — No participants were analyzed for this population at this time point. | 22
  PI-naïve, Week 48; n=20, 49 | 12 | 36
  PI-exp, Week 48; n=0, 40 | NA — No participants were analyzed for this population at this time point. | 19

28. Secondary Outcome: Median Plasma HIV-1 RNA (log10 Copies/mL) at Baseline and Weeks 2, 12, 24, and 48 (Observed Analysis)
Description: Blood samples of participants were collected to assess the decrease in the number of HIV-1 RNA.
Time Frame: Baseline and Weeks 2, 12, 24, and 48
Population: ITT-E Population. In the observed analysis, data are presented for the number of par. still enrolled in the study at a certain time point. The number of par. analyzed represents the sum of the PI-naïve (received <1 week's treatment with a PI) and -experienced (received >1 week prior PI therapy with no more than 3 PIs before trial enrollment) par.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 20 | 88
log10 copies/mL
  PI-naïve, Baseline; n=20, 49 | 5.13 [4.88 to 5.60] | 4.72 [4.27 to 5.20]
  PI-exp, Baseline; n=0, 39 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 4.53 [4.08 to 5.12]
  PI-naïve, Week 2; n=14, 39 | 3.27 [2.65 to 3.89] | 3.06 [2.72 to 3.39]
  PI-exp, Week 2; n=0, 33 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 3.04 [2.66 to 3.49]
  PI-naïve, Week 12; n=19, 46 | 2.03 [1.69 to 2.56] | 1.94 [1.69 to 2.27]
  PI-exp, Week 12; n=0, 34 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 2.20 [1.69 to 3.72]
  PI-naïve, Week 24; n=18, 44 | 1.85 [1.69 to 2.60] | 1.69 [1.69 to 1.95]
  PI-exp, Week 24; n=0, 35 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 1.80 [1.69 to 3.29]
  PI-naïve, Week 48; n=18, 44 | 1.85 [1.69 to 2.60] | 1.69 [1.69 to 1.82]
  PI-exp, Week 48; n=0, 33 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 1.69 [1.69 to 3.51]

29. Secondary Outcome: Median Change From Plasma HIV-1 RNA (log10 Copies/mL) at Weeks 2, 12, 24, and 48 (Observed Analysis)
Description: Blood samples of participants were collected to assess the decrease in the number of HIV-1 RNA. Change from Baseline at Weeks 2, 12, 24, and 48 was calculated as value at Week 2, 12, 24, and 48 minus the value at Baseline.
Time Frame: Baseline and Weeks 2, 12, 24, and 48
Population: as for outcome 28
Measure: Median (Inter-Quartile Range); unit: log10/copies
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 19 | 79
log10/copies
  PI-naïve, Week 2; n=14, 39 | -1.91 [-2.26 to -1.55] | -1.84 [-2.17 to -1.49]
  PI-exp, Week 2; n=0, 32 | NA [NA to NA] — No participants were analyzed for this population at this time point. | -1.58 [-1.97 to -0.70]
  PI-naïve, Week 12; n=19, 46 | -3.04 [-3.21 to -2.70] | -2.77 [-3.22 to -2.28]
  PI-exp, Week 12; n=0, 33 | NA [NA to NA] — No participants were analyzed for this population at this time point. | -2.23 [-2.85 to -1.34]
  PI-naïve, Week 24; n=18, 44 | -3.16 [-3.41 to -2.46] | -2.87 [-3.48 to -2.31]
  PI-exp, Week 24; n=0, 35 | NA [NA to NA] — No participants were analyzed for this population at this time point. | -2.28 [-3.04 to -1.21]
  PI-naïve, Week 48; n=18, 44 | -3.02 [-3.41 to -2.46] | -2.83 [-3.51 to -2.14]
  PI-exp, Week 48; n=0, 33 | NA [NA to NA] — No participants were analyzed for this population at this time point. | -2.14 [-3.04 to -0.92]

30. Secondary Outcome: Number of Participants With at Least a 1.0 log10 HIV-1 RNA Decrease From Baseline at Weeks 2, 12, 24, and 48 (Observed Analysis)
Description: Blood samples of participants were collected to assess the decrease in the number of HIV-1 RNA.
Time Frame: Baseline and Weeks 2, 12, 24, and 48
Population: as for outcome 28
Measure: Number; unit: participants
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 19 | 79
participants
  PI-naïve, Week 2; n=14, 39 | 13 | 35
  PI-exp, Week 2; n=0, 32 | NA — No participants were analyzed for this population at this time point. | 22
  PI-naïve, Week 12; n=19, 46 | 19 | 41
  PI-exp, Week 12; n=0, 33 | NA — No participants were analyzed for this population at this time point. | 26
  PI-naïve, Week 24; n=18, 44 | 18 | 41
  PI-exp, Week 24; n=0, 35 | NA — No participants were analyzed for this population at this time point. | 29
  PI-naïve, Week 48; n=18, 44 | 17 | 40
  PI-exp, Week 48; n=0, 33 | NA — No participants were analyzed for this population at this time point. | 24

31. Secondary Outcome: Cluster of Differentiation Antigen 4 (CD4+) Cell Count at Baseline and at Weeks 2, 12, 24, and 48
Description: Blood samples of participants were collected for the measurement of CD4+ cell count. Observed analysis was used for the summary of proportion endpoints using viral load data. CD4+ cells are white blood cells that are important in fighting infection. HIV infects CD4+ cells, replicates in them, and destroys them. CD4+ cell count provides a measure of the status of the immune system and to what extent it is affected by HIV.
Time Frame: Baseline and Weeks 2, 12, 24, and 48
Population: ITT-E Population. Only those participants contributing data at the indicated time points were analyzed. The number of participants analyzed represents the sum of the PI-naïve (received <1 week's treatment with a PI) and -experienced (received >1 week prior PI therapy with no more than 3 PIs before trial enrollment) participants.
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter (cells/cu mm)
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 19 | 89
Cells per cubic millimeter (cells/cu mm)
  PI-naïve, Baseline; n= 19, 49 | 810 (387.42) [460 to 1000] | 370 (399.39) [200 to 670]
  PI-naïve, Week 2; n= 13, 41 | 820 (370.81) [760 to 1120] | 450 (575.73) [300 to 781]
  PI-naïve, Week 12; n= 19, 46 | 1040 (606.25) [600 to 1440] | 581 (555.52) [310 to 890]
  PI-naïve, Week 24; n= 18, 44 | 1260 (482.92) [1050 to 1640] | 609 (509.24) [341 to 905]
  PI-naïve, Week 48; n= 18, 42 | 1080 (611.28) [570 to 1400] | 670 (568.20) [433 to 910]
  PI-exp, Baseline; n= 0, 40 | NA (0) [NA to NA] — No participants were analyzed for this population at this time point. | 440 (562.00) [220 to 685]
  PI-exp, Week 2; n= 0, 32 | NA (0) [NA to NA] — No participants were analyzed for this population at this time point. | 605 (444.63) [270 to 755]
  PI-exp, Week 12; n= 0, 31 | NA (0) [NA to NA] — No participants were analyzed for this population at this time point. | 720 (379.84) [380 to 870]
  PI-exp, Week 24; n= 0, 34 | NA (0) [NA to NA] — No participants were analyzed for this population at this time point. | 620 (420.62) [370 to 790]
  PI-exp, Week 48; n= 0, 29 | NA (0) [NA to NA] — No participants were analyzed for this population at this time point. | 540 (297.80) [350 to 640]

32. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Weeks 2, 12, 24, and 48
Description: Blood samples of participants were collected for the measurement of CD4+ cell count. Observed analysis was used for the summary of proportion endpoints using viral load data. Change from Baseline was calculated as the value at Weeks 2, 12, 24, and 48 minus the value at Baseline.
Time Frame: Baseline and Weeks 2, 12, 24, and 48
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: cells/cu mm
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 19 | 78
cells/cu mm
  PI-naïve, Week 2; n=13, 41 | 20 [-20 to 180] | 60 [0 to 160]
  PI-naïve, Week 12; n=19, 46 | 170 [50 to 490] | 180 [60 to 269]
  PI-naïve, Week 24; n=18, 44 | 350 [110 to 640] | 184 [53 to 367]
  PI-naïve, Week 48; n=17, 42 | 340 [-40 to 470] | 217 [100 to 398]
  PI-exp, Week 2; n=0, 32 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 90 [2 to 190]
  PI-exp, Week 12; n=0, 31 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 200 [70 to 340]
  PI-exp, Week 24; n=0, 34 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 150 [10 to 260]
  PI-exp, Week 48; n=0, 29 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 180 [0 to 270]

33. Secondary Outcome: Percentage of Total Lymphocytes (TLs) That Are CD4+ Cells at Baseline and Weeks 2, 12, 24, and 48
Description: Blood samples of participants were collected for the measurement of the percentage of total lymphocytes that are CD4+ cells. Observed analysis was used for the summary of proportion endpoints using viral load data.
Time Frame: Baseline and Weeks 2, 12, 24, and 48
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: Percentage of TLs that are CD4+ cells
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 19 | 89
Percentage of TLs that are CD4+ cells
  PI-naïve, Baseline; n=19, 49 | 19 [18 to 27] | 21 [14 to 29]
  PI-naïve, Week 2; n=13, 41 | 24 [22 to 25] | 23 [18 to 30]
  PI-naïve, Week 12; n=19, 46 | 27 [24 to 33] | 25 [17 to 33]
  PI-naïve, Week 24; n=18, 44 | 31 [26 to 34] | 28 [19 to 36]
  PI-naïve, Week 48; n=18, 42 | 32 [27 to 34] | 29 [24 to 36]
  PI-exp, Baseline; n=0, 40 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 24 [11 to 30]
  PI-exp, Week 2; n=0, 32 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 22 [14 to 33]
  PI-exp, Week 12; n=0, 31 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 23 [15 to 34]
  PI-exp, Week 24; n=0, 34 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 23 [17 to 34]
  PI-exp, Week 48; n=0, 29 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 24 [15 to 32]

34. Secondary Outcome: Change From Baseline in the Percentage of Total Lymphocytes (TLs) That Are CD4+ Cells at Weeks 2, 12, 24, and 48
Description: Blood samples of participants were collected for the measurement of the percentage of total lymphocytes that are CD4+ cells. Observed analysis was used for the summary of proportion endpoints using viral load data. Change from Baseline in percentage was calculated as the value at Weeks 2, 12, 24, and 48 minus the value at Baseline.
Time Frame: Baseline and Week 2, 12, 24, 48
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: Percentage of TLs that are CD4+ cells
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 19 | 78
Percentage of TLs that are CD4+ cells
  PI-naïve, Week 2; n=13, 41 | 3 [0 to 5] | 1 [-1 to 4]
  PI-naïve, Week 12; n=19, 46 | 6 [2 to 7] | 5 [1 to 7]
  PI-naïve, Week 24; n=18, 44 | 7 [3 to 11] | 8 [4 to 10]
  PI-naïve, Week 48; n=17, 42 | 8 [4 to 11] | 10 [5 to 14]
  PI-exp, Week 2; n=0, 32 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 2 [0 to 5]
  PI-exp, Week 12; n=0, 31 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 3 [2 to 7]
  PI-exp, Week 24; n=0, 34 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 5 [1 to 8]
  PI-exp, Week 48; n=0, 29 | NA [NA to NA] — No participants were analyzed for this population at this time point. | 6 [2 to 10]

35. Secondary Outcome: Number of Confirmed Virologic Failure Participants (Par.) With Treatment-emergent HIV Genotypic Resistance in Reverse Transcriptase and Protease
Description: A blood sample was drawn for par. failing to respond to therapy, and the mutations present in the virus were identified. For each par., the mutations found at the time of failure were compared with any mutations found in the blood sample at baseline. New International AIDS Society-USA defined resistance mutations that developed at the time of failure were tabulated by drug class. VF, virologic failure; NRTI, nucleoside reverse transcriptase inhibitor; NNRTI, non-nucleoside reverse transcriptase inhibitor; PI, protease inhibitor. Par. are grouped by study arm and prior therapy experience.
Time Frame: Week 48
Population: VF: par. with failure to achieve plasma HIV-RNA <400 copies/mL by Week 24; or confirmed HIV-RNA rebound to >=400 copies/mL any time after achieving plasma HIV-RNA <400 copies/mL and had evaluable viral isolate genotypic and/or phenotypic data. Only par. contributing viral genotype at both baseline and the indicated time of VF points were evaluable.
Measure: Number; unit: participants
Groups:
- ART-Naïve, FPV Treatment Group: Human immunodeficiency virus type 1 (HIV-1)-infected, antiretroviral-naive pediatric participants, 2 to <6 years old, receiving fosamprenavir (FPV) oral suspension 30-40 milligrams per kilogram (mg/kg) twice a day (BID)
- ART-Naïve, FPV/RTV Treatment Group: HIV-1-infected, antiretroviral-naïve pediatric participants, 2 to 18 years old, receiving FPV boosted with ritonavir (FPV/RTV) BID
- PI Naïve, ART Experienced, FPV/RTV Treatment Group: HIV-1-infected, antiretroviral-experienced but PI-naïve pediatric participants, 2 to 18 years old, receiving FPV boosted with ritonavir (FPV/RTV) BID
- PI Experienced, ART Experienced, FPV/RTV Treatment Group: HIV-1-infected, PI-experienced pediatric participants, 2 to 18 years old, receiving FPV boosted with ritonavir (FPV/RTV) BID
Arm/Group | ART-Naïve, FPV Treatment Group | ART-Naïve, FPV/RTV Treatment Group | PI Naïve, ART Experienced, FPV/RTV Treatment Group | PI Experienced, ART Experienced, FPV/RTV Treatment Group
Number analyzed (Participants) | 3 | 1 | 3 | 8
participants
  Any HIV NRTI Mutation | 3 | 0 | 0 | 1
  HIV NRTI mutation M184V | 3 | 0 | 0 | 1
  Any HIV NNRTI Mutation | 0 | 0 | 0 | 1
  HIV NNRTI Mutation V179D/E | 0 | 0 | 0 | 1
  Any HIV Major PI Mutations | 2 | 0 | 1 | 1
  HIV Major PI Mutation M46M/I | 0 | 0 | 1 | 0
  HIV Major PI Mutation M46M/L | 1 | 0 | 0 | 0
  HIV Major PI Mutation I50I/V | 1 | 0 | 1 | 1
  HIV Major PI Mutation I54I/L | 1 | 0 | 0 | 0
  HIV Major PI Mutation I54I/M | 0 | 0 | 0 | 1
  HIV Major PI Mutation I54I/M/V | 0 | 0 | 1 | 0
  HIV Major PI Mutation Q58Q/E | 1 | 0 | 0 | 0
  HIV Major PI Mutation V82A/V | 1 | 0 | 0 | 0
  HIV Major PI Mutation V82F/I | 0 | 0 | 0 | 1
  HIV Major PI Mutation I84I/V | 0 | 0 | 1 | 0
  Any Minor HIV PI Mutations | 2 | 0 | 1 | 1
  Minor HIV PI Mutation L10L/F | 0 | 0 | 1 | 0
  Minor HIV PI Mutation K20K/R | 1 | 0 | 0 | 0
  Minor HIV PI Mutation L33L/F | 1 | 0 | 1 | 0
  Minor HIV PI Mutation K43K/T | 0 | 0 | 0 | 1
  Minor HIV PI Mutation F53F/L | 1 | 0 | 0 | 0
  Minor HIV PI Mutation F53L | 1 | 0 | 0 | 0
  Minor HIV PI Mutation I62I/V | 0 | 0 | 1 | 0
  Minor HIV PI Mutation A71I/V | 0 | 0 | 1 | 0
  Minor HIV PI Mutation I85I/V | 0 | 0 | 1 | 1

36. Secondary Outcome: Number of Confirmed Virologic Failure Participants (Par.) Since the Week 48 Analysis With Treatment-emergent HIV Genotypic Resistance in Reverse Transcriptase and Protease
Description: A blood sample was drawn for par. remaining in the study after Week 48 and failing to respond to therapy, and the mutations present in the virus were identified. For each par., the mutations found at the time of failure were compared with any mutations found in the blood sample at baseline. New International AIDS Society-USA defined resistance mutations that developed at the time of failure were tabulated by drug class. VF, virologic failure; NRTI, nucleoside reverse transcriptase inhibitor; NNRTI, non-nucleoside reverse transcriptase inhibitor; PI, protease inhibitor. Par. are grouped by study arm and prior therapy experience.
Time Frame: After Week 48 through Week 240
Population: as for outcome 35
Measure: Number; unit: Participants
Arm/Group | ART-Naïve, FPV Treatment Group | ART-Naïve, FPV/RTV Treatment Group | PI Naïve, ART Experienced, FPV/RTV Treatment Group | PI Experienced, ART Experienced, FPV/RTV Treatment Group
Number analyzed (Participants) | 1 | 1 | 0 | 5
Participants
  Any HIV NRTI Mutation | 1 | 1 |  | 2
  HIV NRTI mutation M41L | 0 | 0 |  | 1
  HIV NRTI mutation M184I | 0 | 1 |  | 0
  HIV NRTI mutation M184V | 1 | 0 |  | 2
  HIV NRTI mutation T215S/Y | 0 | 0 |  | 1
  Any Major HIV NNRTI Mutation | 0 | 0 |  | 1
  HIV NNRTI Mutation K103N | 0 | 0 |  | 1
  Any Minor HIV NNRTI Mutation | 0 | 0 |  | 0
  HIV NNRTI Mutation V179D/E | 0 | 0 |  | 0
  Any HIV Major PI Mutations | 1 | 0 |  | 1
  HIV Major PI Mutation V32I | 0 | 0 |  | 1
  HIV Major PI Mutation M46L | 1 | 0 |  | 0
  HIV Major PI Mutation I47IV | 0 | 0 |  | 1
  HIV Major PI Mutation T74P | 1 | 0 |  | 0
  HIV Major PI Mutation I84I/V | 0 | 0 |  | 0
  Any Minor HIV PI Mutations | 1 | 0 |  | 2
  Minor HIV PI Mutation L10F | 1 | 0 |  | 0
  Minor HIV PI Mutation L33F | 0 | 0 |  | 1
  Minor HIV PI Mutation I62I/V | 0 | 0 |  | 1
  Minor HIV PI Mutation I85V | 1 | 0 |  | 0

37. Secondary Outcome: Number of Confirmed Virologic Failure Participants (Par.) With Treatment-emergent Reductions in Drug Susceptibility (DS)
Description: A blood sample was drawn for par. failing to respond to therapy, and changes in DS for HIV isolated from the par. for each drug used in the study were assessed. The changes in DS detected by phenotypic assay in virus from the sample collected at the time of failure was compared with DS in the virus from the blood sample at baseline. Par. are grouped by study arm and prior therapy experience. DS is the state of HIV being susceptible to the antiretroviral agent (the virus can be inhibited by the drug). Reduced DS (i.e., HIV is resistant to the antiretroviral agent) can lead to treatment failure.
Time Frame: Baseline through 48 Weeks
Population: VF: par. with failure to achieve plasma HIV-RNA <400 copies/mL by Week 24; or confirmed HIV-RNA rebound to >=400 copies/mL any time after achieving plasma HIV-RNA <400 copies/mL and had evaluable viral isolate genotypic and/or phenotypic data. Only par. contributing viral phenotype at both baseline and the indicated time of VF points were evaluable
Measure: Number; unit: participants
Groups:
- PI Naïve, ART-experienced, FPV/RTV Treatment Group: HIV-1-infected, antiretroviral-experienced but PI- pediatric participants, 2 to 18 years old, receiving FPV boosted with ritonavir (FPV/RTV) BID
- PI-experienced, ART-experienced FPV/RTV Treatment Group: HIV-1-infected, PI-experienced pediatric participants, 2 to 18 years old, receiving FPV boosted with ritonavir (FPV/RTV) BID
Arm/Group | ART-Naïve, FPV Treatment Group | ART-Naïve, FPV/RTV Treatment Group | PI Naïve, ART-experienced, FPV/RTV Treatment Group | PI-experienced, ART-experienced FPV/RTV Treatment Group
Number analyzed (Participants) | 3 | 1 | 3 | 8
participants
  Any NRTI | 3 | 0 | 0 | 2
  Abacavir | 1 | 0 | 0 | 0
  Didanosine | 3 | 0 | 0 | 1
  Emtricitabine | 3 | 0 | 0 | 1
  Lamivudine | 3 | 0 | 0 | 1
  Any NNRTI | 0 | 0 | 0 | 0
  Any PI | 2 | 0 | 1 | 1
  Unboosted Fosamprenavir | 2 | NA — These participants took RTV-boosted FPV. | NA — These participants took RTV-boosted FPV. | NA — These participants took RTV-boosted FPV.
  Ritonavir- boosted Fosamprenavir | NA — These participants took unboosted FPV. | 0 | 1 | 1
  Ritonavir | 2 | 0 | 0 | 0

38. Secondary Outcome: Number of Confirmed Virologic Failure Participants (Par.) Since the Week 48 Analysis With Treatment-emergent Reductions in Drug Susceptibility (DS)
Description: A blood sample was drawn for par. remaining in the study after Week 48 and failing to respond to therapy, and changes in DS for HIV isolated from the par. for each drug used in the study were assessed. The changes in DS detected by phenotypic assay in virus from the sample collected at the time of failure was compared with DS in the virus from the blood sample at baseline. Par. are grouped by study arm and prior therapy experience. DS is the state of HIV being susceptible to the antiretroviral agent (the virus can be inhibited by the drug). Reduced DS (i.e., HIV is resistant to the antiretroviral agent) can lead to treatment failure.
Time Frame: Week 60 through Week 240
Population: as for outcome 37
Measure: Number; unit: Participants
Arm/Group | ART-Naïve, FPV Treatment Group | ART-Naïve, FPV/RTV Treatment Group | PI Naïve, ART-experienced, FPV/RTV Treatment Group | PI-experienced, ART-experienced FPV/RTV Treatment Group
Number analyzed (Participants) | 1 | 1 | 0 | 5
Participants
  Any NRTI | 1 | 1 |  | 3
  Abacavir | 0 | 0 |  | 1
  Didanosine | 0 | 1 |  | 3
  Emtricitabine | 1 | 1 |  | 3
  Lamivudine | 1 | 1 |  | 2
  Zidovudine | 0 | 0 |  | 1
  Any NNRTI | 0 | 0 |  | 1
  Delaviridine | 0 | 0 |  | 1
  Efavirenz | 0 | 0 |  | 1
  Nevirapine | 0 | 0 |  | 1
  Any PI | 1 | 1 |  | 3
  Unboosted Fosamprenavir | 1 | NA — These participants took RTV-boosted FPV. |  | NA — These participants took RTV-boosted FPV
  Ritonavir- boosted Fosamprenavir | NA — These participants took unboosted FPV. | 0 |  | 1
  Nelfinavir | 0 | 1 |  | 0
  Tipranavir | 0 | 0 |  | 1

39. Secondary Outcome: Number of Participants Reporting Perfect Adherence Over the 3 Days Prior to the Study Visits at Weeks 2, 12, 24, and 48 as Assessed by Study Coordinator Using the Pediatric AIDS Clinical Trials Group (PACTG) Adherence Questionnaire
Description: The PACTG Adherence Questionnaire records individual study drugs, the expected number of doses/24 hour period, and the number of doses missed in the 3 days prior to the study visit. Responses were summarized by age cohort, study drug, treatment regimen, and visit for exploratory analysis only.
Time Frame: Weeks 2, 12, 24, and 48
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 17 | 59
participants
  Week 2, Total Population; n= 17, 59 | 15 | 49
  Week 2, 2 to <6 years (yrs); n= 17, 16 | 15 | 15
  Week 2, 6 to <12 yrs; n= 0, 25 | NA — No participants were analyzed for this population at this time point. | 22
  Week 2, 12 to 18 yrs; n= 0, 18 | NA — No participants were analyzed for this population at this time point. | 12
  Week 12, Total Population; n= 16, 55 | 15 | 45
  Week 12, 2 to <6 yrs; n= 16, 16 | 15 | 14
  Week 12, 6 to <12 yrs; n= 0, 24 | NA — No participants were analyzed for this population at this time point. | 20
  Week 12, 12 to 18 yrs; n= 0, 15 | NA — No participants were analyzed for this population at this time point. | 11
  Week 24, Total Population; n= 16, 54 | 16 | 43
  Week 24, 2 to <6 yrs; n= 16, 14 | 16 | 11
  Week 24, 6 to <12 yrs; n= 0, 24 | NA — No participants were analyzed for this population at this time point. | 23
  Week 24, 12 to 18 yrs; n= 0, 16 | NA — No participants were analyzed for this population at this time point. | 9
  Week 48, Total Population; n= 15, 53 | 13 | 42
  Week 48, 2 to <6 yrs; n= 15, 14 | 13 | 13
  Week 48, 6 to <12 yrs; n= 0, 23 | NA — No participants were analyzed for this population at this time point. | 20
  Week 48, 12 to 18 yrs; n= 0, 16 | NA — No participants were analyzed for this population at this time point. | 9

40. Secondary Outcome: Correlation Between Plasma APV Exposure and Plasma vRNA, CD4+ Cell Counts, and the Occurrence of Adverse Events
Description: No formal analysis has been performed or is planned to correlate plasma APV PK with efficacy and safety outcomes.
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | FPV Treatment Group | FPV/RTV Treatment Group
Serious Adverse Events (participants affected / at risk) | 5/20 | 13/89
Other Adverse Events (participants affected / at risk) | 18/20 | 74/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FPV Treatment Group (N=20) | FPV/RTV Treatment Group (N=89)
Drug hypersensitivity (Immune system disorders) | 3 | 6
Pneumonia (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1
Measles (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FPV Treatment Group (N=20) | FPV/RTV Treatment Group (N=89)
Vomiting (Gastrointestinal disorders) | 12 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 33
Diarrhea (Gastrointestinal disorders) | 2 | 26
Upper respiratory tract infection (Infections and infestations) | 3 | 20
Pyrexia (General disorders) | 1 | 19
Nasopharyngitis (Infections and infestations) | 1 | 16
Respiratory tract infection (Infections and infestations) | 12 | 4
Rhinitis (Infections and infestations) | 2 | 15
Bronchitis (Infections and infestations) | 3 | 12
Ear infection (Infections and infestations) | 3 | 11
Headache (Nervous system disorders) | 0 | 14
Rash (Skin and subcutaneous tissue disorders) | 0 | 14
Nausea (Gastrointestinal disorders) | 1 | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 10
Otitis media (Infections and infestations) | 0 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Pharyngitis (Infections and infestations) | 1 | 8
Conjunctivitis (Eye disorders) | 0 | 8
Gasrtroenteritis (Infections and infestations) | 0 | 7
Abdominal pain (Gastrointestinal disorders) | 0 | 7
Ear pain (Ear and labyrinth disorders) | 0 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Eczema (Skin and subcutaneous tissue disorders) | 1 | 5
Tonsillitis (Infections and infestations) | 1 | 6
Dental caries (Gastrointestinal disorders) | 0 | 6
Tinea capitis (Infections and infestations) | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.